CLINICAL TRIAL: NCT05343559
Title: The Influence of a Mask on the First Impressions Projected and Attractiveness Levels of Smiling Individuals
Brief Title: First Impressions and Attractiveness Levels of Smiling Individuals With and Without a Mask
Status: Completed | Type: Observational
Sponsor: DeNova Research (Other)
Responsible Party: Principal Investigator, Steven H. Dayan, MD, DeNova Research
Other Study IDs: Smile-2022
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: First Impressions; Attractiveness
Keywords: attractiveness; first impressions; smiling; mask; masking; rating
MeSH Terms: conditions — Smiling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluation on the effects of smiling on first impressions and attractiveness with and without wearing a facial surgical mask.

ELIGIBILITY:
Inclusion Criteria:

1. Models who are males and females of ages 21-39.
2. Live and random raters who are males and females of ages 18-39.
3. Models and raters that understand the purpose and aspects of the study, freely sign the consent and complete the required visit.
4. Models and raters must all be able to understand English fluently.

Exclusion Criteria:

1. Model participants younger than 21 or older than 40 will not be included.
2. Live and random rater participants younger than 18 and older than 40 will not be included.
3. Models with unusual hair styles or colors
4. Facial piercing other than ears
5. Facial and/or neck scaring or tattooing
6. Models and raters that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required visit will also be excluded.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — 4 models identifying as female and 4 models identifying as male
Study Population: Inclusion Criteria:
  1. Models who are males and females of ages 21-39.
  2. Live and random raters who are males and females of ages 18-39.
  3. Models and raters that understand the purpose and aspects of the study, freely sign the consent and complete the required visit.
  4. Models and raters must all be able to understand English fluently.
  Exclusion Criteria:
  1. Model participants younger than 21 or older than 40 will not be included.
  2. Live and random rater participants younger than 18 and older than 40 will not be included.
  3. Models with unusual hair styles or colors
  4. Facial piercing other than ears
  5. Facial and/or neck scaring or tattooing
  6. Models and raters that do not understand the purpose and aspects of the study, do not sign the consent and do not complete the required visit will also be excluded.
Sampling Method: Probability Sample
Enrollment: 808 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of smiling on first impressions with and without wearing a mask | 8 weeks
  First impression questionnaire (FIQ)

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States